CLINICAL TRIAL: NCT05318443
Title: A Randomized, Double-blind, Parallel-controlled Study Comparing the Efficacy and Safety of Recombinant Anti-VEGF Humanized Monoclonal Antibody Injection (SIBP04) and Bevacizumab Injection (Avastin) in Combination With Paclitaxel and Carboplatin Respectively in Patients With Advanced, Metastatic or Recurrent Non-squamous Non-small Cell Lung Cancer.
Brief Title: A Study Exploring Efficacy of SIBP04 in Subjects With Non-squamous Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Institute Of Biological Products (Industry)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIBP04-02
Record Dates: First submitted 2022-03-22; First posted 2022-04-08 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-09

CONDITIONS: Non-squamous Non-small-cell Lung Cancer
Keywords: Non-squamous Non-small-cell Lung Cancer; Efficacy; Safety; Tolerability; Pharmacokinetics
MeSH Terms: interventions — Bevacizumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, parallel-controlled, multicenter Phase III clinical study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): SIBP04 & Paclitaxel & Carboplatin
  Interventions: Drug: SIBP04; Drug: Paclitaxel; Drug: Carboplatin
- Control group (Active Comparator): Avastin & Paclitaxel & Carboplatin
  Interventions: Drug: Avastin; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: SIBP04 — SIBP04, 15mg/kg, intravenous infusion, the first intravenous infusion 90min (+10min), 3 weeks/cycle, administered on the first day of each treatment cycle.
  Arms: Experimental
Drug: Avastin — Avastin, 15mg/kg, intravenous infusion, the first intravenous infusion 90min (+10min), 3 weeks/cycle, administered on the first day of each treatment cycle.
  Arms: Control group
Drug: Paclitaxel — Paclitaxel, 175mg/m2, intravenous infusion, every 3 weeks/cycle, administered on the first day of each treatment cycle.
Drug: Carboplatin — Carboplatin, AUC=5.0, (upper limit 800mg), intravenous infusion, 3 weeks/cycle, administered on the first day of each treatment cycle.

SUMMARY:
This trial is a randomized, double-blind, parallel-controlled, multicenter phase III clinical study. To evaluate the clinical efficacy of SIBP04 in patients with locally advanced, metastatic or recurrent non-squamous non-small cell lung cancer.

DETAILED DESCRIPTION:
This trial is a randomized, double-blind, parallel-controlled, multicenter phase III clinical study. The study was divided into three stages: screening stage, treatment stage (combined chemotherapy stage, single drug maintenance treatment stage, visit after treatment) and follow-up stage (survival follow-up after disease progression). To evaluate the safety, tolerability, pharmacokinetics and clinical efficacy of SIBP04 in patients with locally advanced, metastatic or recurrent non-squamous non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* The subjects voluntarily joined the trial and signed the informed consent form;
* Age≥18 years old and≤75 years old (subject to the date of signing the informed consent form), male or female;
* Non-squamous non-small cell lung cancer confirmed by histology or cytology (excluding sputum cytology), and according to the International Association for the Study of Lung Cancer (IASLC) eighth edition staging criteria, evaluated as stage IIIB-IV inoperable treatment or locally advanced, recurrent or metastatic subjects who cannot receive radical radiotherapy or refuse radical radiotherapy; if there are multiple tumor components, they should be classified according to their main cell types;
* EGFR, ALK, ROS-1 positive patients can be enrolled voluntarily, and the subjects need to provide the test results report of the above genes (If the subject fails to provide the EGFR, ALK, ROS-1 gene test report, he or she must provide tissue sections or tumor specimens for testing in this research center or a tertiary hospital. When the driver gene is unknown, the investigator and the subject jointly decide whether to join the group);
* At least one evaluable target lesion confirmed by imaging (evaluated according to RECIST 1.1 criteria);
* ECOG PS score is 0-1;
* Expected survival time ≥ 6 months;
* No systematic anti-tumor treatment for locally advanced or metastatic non-squamous non-small cell lung cancer [Subjects can be enrolled if they receive adjuvant therapy after completing curative treatment for early-stage non-small cell lung cancer, but have disease recurrence. In this case, the end time of adjuvant therapy is required to be more than 6 months after the first administration of this study, and the various toxic reactions caused by adjuvant therapy have recovered (judged by CTCAE 5.0 standard ≤ grade 1, except for alopecia ) or a new lesion appeared 6 months after the end of radical radiotherapy in stage IIIB patients]
* Laboratory results at screening:

Blood routine: white blood cell count≥3.5×109/L, absolute value of neutrophil ≥1.5×109/L, platelet count ≥100×109/L, hemoglobin ≥100g/L; Liver function: total bilirubin ≤1.5× upper limit of normal (ULN); subjects without liver metastases had alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN; liver Metastatic subjects with ALT and AST ≤ 5×ULN; Renal function: Serum creatinine ≤1.5×ULN or creatinine clearance ≥ 55mL/min, and urine routine test results show urine protein <2+, for subjects whose urine routine test shows urine protein ≥2+ at baseline, 24 hours urine collection should be performed and protein content in urine <1.0g within 24 hours; Coagulation function: International Normalized Ratio (INR) ≤1.5, and Activated Partial Thromboplastin Time (APTT) ≤1.5×ULN;

* Female subjects of childbearing age, male subjects and male subjects' partners agree to use reliable contraceptive measures from the time of signing the informed consent to 6 months after the end of the last trial drug infusion (such as abstinence, or physical contraception, or hormonal contraception, etc.);
* Subjects need to communicate well with the investigator, and be able to follow the visit, treatment, laboratory examination and other relevant regulations.

Exclusion Criteria:

* Subjects with non-small cell lung cancer of other pathological histological types [including squamous cell carcinoma, mixed non-small cell and small cell lung cancer, and lung adenosquamous carcinoma with squamous cell carcinoma predominant];
* Malignant tumors other than lung cancer within 5 years, excluding cured cervical carcinoma in situ, skin basal cell or squamous cell skin cancer, local prostate cancer after radical resection, and breast ductal carcinoma in situ after radical resection, etc. ;
* Left ventricular ejection fraction (LVEF) < 50% by color Doppler echocardiography;
* Imaging examination at the screening stage show that the tumor approaches, surrounds, or invades the lumen of a large vessel (eg, the pulmonary artery or superior vena cava);
* Subjects with high suspicion of idiopathic pulmonary fibrosis, organizing pneumonia, drug-related pneumonia, idiopathic pneumonia, active pneumonia or active pulmonary tuberculosis by chest imaging examination during the screening stage;
* Previous history of hypertensive crisis, hypertensive encephalopathy; or uncontrolled hypertension (systolic blood pressure>150mmHg, and/or diastolic blood pressure>100mmHg);
* Any unstable systemic disease within 6 months prior to randomization: Including but not limited to cerebrovascular accident or transient ischemic attack, unstable angina pectoris, myocardial infarction, congestive heart failure [New York Heart Association (NYHA) grade ≥ grade II], severe arrhythmia requiring drug treatment, etc.;
* There are serious unhealed wounds or fractures, or major surgery (including thoracotomy, or major surgery is expected during the study period) within 28 days before randomization; For major surgery, refer to the 3rd and 4th grade surgery stipulated in the "Administrative Measures for the Classification of Surgery in Medical Institutions (Trial)";
* Subjects who have undergone minor surgery within 48 hours before randomization, and who are judged by the investigator to have a bleeding tendency;
* Subjects who have a history of chest radiotherapy within 28 days before randomization, or those who have received palliative radiotherapy for bone metastases within 14 days before randomization;
* History of the following within 6 months before randomization: peptic ulcer, gastrointestinal perforation, erosive esophagitis or gastritis, inflammatory bowel disease or diverticulitis, abdominal fistula, or intra-abdominal abscess;
* Definite diagnosis of tracheoesophageal fistula;
* Bleeding tendency, high bleeding risk, or coagulation disorder, including history of hemoptysis within 3 months before screening (single hemoptysis ≥ 2.5 ml bright red blood),or recently (≤10 days from first dose of study drug) full-dose oral or parenteral anticoagulants or thrombolytics or aspirin (>325 mg/day) or other non-steroidal anti-inflammatory drugs that inhibit platelet function; or have undergone surgery before, and the investigator judges that they have bleeding tendency;
* Subjects with known central nervous system metastases (except for the subjects with asymptomatic brain metastases and whose symptoms were controlled after treatment and stable within 1 month before randomization);
* Serious infection (including but not limited to infection requiring hospitalization, bacteremia, severe pneumonia, etc.) occurred within 28 days before randomization;
* A history of vascular disease requiring surgical repair within 6 months prior to randomization, such as aortic aneurysm or arterial thrombosis;
* Known to be allergic to SIBP04, Avastin®, Paclitaxel, Carboplatin injection or their excipients;
* Known history of autoimmune disease, allergic disease or allergic constitution (allergic to two or more foods and drugs);
* Received any other experimental drug treatment or participated in another interventional clinical trial within 3 months before screening;
* In the screening stage, Hepatitis B surface antigen was positive, and the level of hepatitis B virus DNA (HBV-DNA) in peripheral blood was higher than the reference value or lower limit of detection method; Hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody or Treponema pallidum antibody test was positive;
* Pregnant or lactating women or women preparing to be pregnant or lactating during the study period, or with a positive pregnancy test result at screening stage or baseline;
* Uncontrollable pericardial effusion, abdominal cavity, pleural effusion and other third space effusion within 14 days before randomization, and the investigator judges that they are not suitable for this study;
* Other circumstances determined by the investigator as unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 512 (Actual)
Dates: Start 2020-04-17 (Actual); Primary Completion 2022-12-26 (Actual); Study Completion 2023-01-12 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to 18th week.
  ORR is defined as the best ORR from the first medication to the 18th week, initially evaluated by the investigator, and finally evaluated by a third-party independent blinded imaging, including cases of complete response (CR) and partial response (PR).

SECONDARY OUTCOMES:
Progression-free survival(PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 18 weeks.
  PFS is defined as the time between randomization and disease progression or death(The date when event happened first).
Overall survival (OS) | From date of randomization until the date of event-occurring or last visit, assessed up to 30 weeks.
  OS is defined as the time between randomization and patient death from all causes, with the date of last contact as the cut-off date if the patient is lost to follow-up.
Duration of response (DOR) | From date of the first evaluation of a tumor as CR or PR until the date of the first evaluation of a patient's state as disease progression or death, assessed up to 30 weeks.
  DOR is defined as the time from the first evaluation of a tumor as CR or PR to the first evaluation of disease progression or death.
Disease control rate (DCR) | up to 18th week.
  DCR was defined as the percentage of the total evaluable cases with remission or disease stabilization after treatment (That is, cases of CR, PR and stable disease(SD)).

OTHER OUTCOMES:
The number of adverse events (AE) | The last 1 day of 18th weeks after randomization.
  Total number of any spontaneously reported and all directly observed adverse events.
The number of serious adverse events (SAE) | The last 1 day of 30th weeks after randomization.
  That is serious adverse events, any serious adverse events that occurred to the subject during the study period.
The incidence of anti-drug antibodies(ADAs) | The last 1 day of 18th weeks after randomization.
  Evaluate the immunogenicity of the SIBP04 group and the bevacizumab group.
The titer of ADAs | The last 1 day of 18th weeks after randomization.
  Evaluate the immunogenicity of the SIBP04 group and the bevacizumab group.
The incidence of neutralizing antibodies (NAbs) | The last 1 day of 18th weeks after randomization.
  Evaluate the immunogenicity of the SIBP04 group and the bevacizumab group.
The trough concentration | The last 1 day of 18th weeks after randomization.
  The trough concentration is a pharmacokinetic evaluation index.

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, Doctor, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Aidong Qu, Master, Study Director — Co., Ltd Shanghai Institute Of Biological Products
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shi Y, Bi M, Li Q, Wang G, Chen J, Li M, Shi J, Mei J, Ji Y, Xia Q, Feng Y, Xu S, Zhang T, Gao X, Tang S, Weng J, Cao Z, Wu H, Ren X, Xie H, Liu H, Liu Q, Yin X, Luo X, Chen J, Zhang H, Guo Z, Ding C, Jin X, Sun R, Yang S. Efficacy and safety of bevacizumab biosimilar SIBP04 compared with bevacizumab (Avastin(R)) as first-line treatment for locally advanced or metastatic non-squamous non-small-cell lung cancer: A randomized, double-blind, phase 3 trial. Cancer Pathog Ther. 2025 Jan 6;3(4):337-345. doi: 10.1016/j.cpt.2025.01.001. eCollection 2025 Jul. PMID 40697509
- [Derived] Qu A, Zhang S, Zou H, Li S, Chen D, Zhang Y, Li S, Zhang H, Yang J, Yang Y, Huang Y, Li X, Zhang Y. Outcome benefits of bevacizumab biosimilar (SIBP04) combined with carboplatin and paclitaxel in advanced non-squamous non-small-cell lung cancer patients with EGFR mutation: subgroup analysis of a prospective, randomized phase III clinical trial. J Cancer Res Clin Oncol. 2023 Nov;149(14):12713-12721. doi: 10.1007/s00432-023-05103-4. Epub 2023 Jul 15. PMID 37452849